CLINICAL TRIAL: NCT00261742
Title: Comparative Trial of Oral Penicillin Versus Cefuroxim for Treatment of Perianal Dermatitis - an Open, Randomized, Controlled Trial
Brief Title: Comparative Trial of Oral Penicillin Versus Cefuroxim for Treatment of Perianal Streptococcal Dermatitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214/05
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Streptococcal Infections
Keywords: perianal; dermatitis; streptococcus pyogenes
MeSH Terms: conditions — Streptococcal Infections; Dermatitis

INTERVENTIONS:
Drug: Penicillin versus cefuroxim per os

SUMMARY:
The goal of the study is to investigate, which of two antibiotic treatments - oral penicillin for 10 days or oral cefuroxim for 7 days - is more successful for patients (1-16 years of age) with perianal dermatitis caused by group A beta-hemolytic streptococci.

DETAILED DESCRIPTION:
The goal of the study is to investigate, which of two antibiotic treatments - oral penicillin for 10 days or oral cefuroxim for 7 days - is more successful for patients (1-16 years of age) with perianal dermatitis caused by group A beta-hemolytic streptococci (GABHS). Diagnosis is based on positive perianal culture for GABHS. Informed consent will be obtained.

The study will be performed in the region of Basel, Switzerland, in private practices of pediatricians, general practitioners, and selected pediatric dermatologists as well as in the out-patient departments of the University Children's Hospital Basel and the department for dermatology of the University of Basel.

Patients (or their parents) will fill in a daily diary on signs and symptoms of disease; furthermore, clinical investigations (inspection of the site of infection) will be performed on enrollment (Day 1), Day 3, and at the end of treatment (Day 10).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age 1-16 years
* typical clinical symptoms for perianal dermatitis
* positive perianal culture for GABHS

Exclusion Criteria:

* antibiotic treatment in previous 14 days
* immunodeficiency
* penicillin allergy
* cephalosporin allergy
* further bacterial infections

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194
Dates: Start 2005-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Resolving signs and symptoms of perianal dermatitis

SECONDARY OUTCOMES:
microbiological cure (= negative culture for GABHS) at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Heininger, MD, Principal Investigator — University Children's Hospital Basel; Urs B Schaad, MD, Study Director — University Children's Hospital Basel
Locations (1):
- University Children's Hospital, Basel, Switzerland

REFERENCES:
- [Background] Landolt M, Heininger U. [Prevalence of perianal streptococcal dermatitis in children and adolescents]. Praxis (Bern 1994). 2005 Sep 21;94(38):1467-71. doi: 10.1024/0369-8394.94.38.1467. German. PMID 16209362